CLINICAL TRIAL: NCT00000485
Title: Hypertension Detection and Follow-up Program (HDFP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 4
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2005-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diuretics; Antihypertensive Agents

INTERVENTIONS:
Drug: diuretics
Drug: antihypertensive agents

SUMMARY:
To determine the effectiveness of systematic, sustained, antihypertensive therapy in reducing morbidity and mortality from hypertension in a wide spectrum of persons with elevated blood pressure in 14 communities. During its course, the trial also obtained a direct measure of the prevalence, severity, and treatment status of representative white and black populations with high blood pressure in these 14 communities, and obtained an estimate of the extent of attainable reduction of complications of high blood pressure by an organized screening and blood pressure management program.

DETAILED DESCRIPTION:
BACKGROUND:

Published data from the Veterans Administration Cooperative Study of Hypertension demonstrated that reduction in morbidity and mortality could be attained by treating men with fixed diastolic blood pressure over 105 mm Hg. Similar trends occurred for those with fixed diastolic blood pressure between 90 and 104 mm Hg. Results and current trends from other studies supported these findings. However, prior to inception of the Hypertension Detection and Follow-up Program (HDFP), it was not known whether benefits from antihypertensive therapy applied to all hypertensives in the general population and whether making use of existing medical knowledge could significantly reduce morbidity and mortality from hypertension in communities.

Recognizing this need, NHLBI initiated the pilot activities of the HDFP to characterize significant operational, socioeconomic, and motivational factors that would influence the acceptance of antihypertensive therapy in the defined populations within which the controlled clinical trial would take place and to obtain baseline information necessary to the undertaking of the clinical trial, which was to determine whether a practical, intensive, and antihypertensive program could significantly reduce morbidity and mortality in hypertensives in the general population.

The planning of the trial, including the development of a protocol and manual of operations, began in 1971. Between February 1973 and May 1974, 158,906 persons were screened for high blood pressure in 14 communities. A total of 10,940 hypertensive participants were randomized.

The primary hypothesis tested by the trial was that intensive blood pressure control under stepped care for five years could significantly reduce mortality compared with that under referred-care. Stepped-care was the method of treatment in HDFP clinics in which a diuretic was given initially and additional antihypertensive agents were added in a time-structured, stepwise fashion until goal blood pressure was achieved. Referred-care represented referral to private physicians and other community sources of care. Participating in this study were 14 clinical centers, a coordinating center, ECG center, central laboratory, and monitoring laboratory.

The clinical phase of the trial ended in May 1982. The project was extended into 1983 in order to continue the surveillance of mortality and blood pressure control.

DESIGN NARRATIVE:

The trial was a randomized, non-blind, fixed sample trial with single intervention and control groups. The intervention group received stepped care from the clinical trial clinics (see Background, below), while those in the control group were referred to their own physicians. Each community contributed both stepped-care and referred-care participants, but for analysis purposes, the groups were pooled into two groups. The primary endpoint was mortality. The effects of stepped- vs. referred-care were also assessed on intermediate and secondary factors, including nosologic codes of specific causes of mortality, nonfatal myocardial infarction, stroke, hypertensive heart disease, and EKG abnormalities.

ELIGIBILITY:
Men and women, ages 30-69. Hypertension. Diastolic blood pressure home readings and clinic readings equal to or above 95 mm Hg and 90 mm Hg, respectively.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1971-05; Study Completion 1982-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Hawkins — University of Texas

REFERENCES:
- [Background] Remington RD On behalf of the HDFP Cooperative Group: The Hypertension Detection and Follow-up Program. Inserm, 21:185-194, 1973.
- [Background] Mild hypertensives in the hypertension detection and follow-up program. The Hypertension Detection and Follow-up Cooperative Group. Ann N Y Acad Sci. 1978 Mar 30;304:254-66. doi: 10.1111/j.1749-6632.1978.tb25603.x. No abstract available. PMID 280231
- [Background] Patient participation in a hypertension control program. Hypertension Detection and Follow-up Program Cooperative Group. JAMA. 1978 Apr 14;239(15):1507-14. PMID 633560
- [Background] Variability of blood pressure and the results of screening in the hypertension detection and follow-up program. J Chronic Dis. 1978;31(11):651-67. doi: 10.1016/0021-9681(78)90069-3. No abstract available. PMID 730822
- [Background] Hypertension and Education. Journal of the American Dietetic Association, 72 (4):377, April l978. (Summary of Mainstream Paper #5A.)
- [Background] Blood Pressure Studies in l4 Communities: A Two-Stage Screen for Hypertension. l978 Year Book of Cardiology: 355-57 (Summary of Mainstream Paper #2.)
- [Background] Therapeutic control of blood pressure in the Hypertension Detection and Follow-up Program. Hypertension Detection and Follow-up Program Cooperative Group. Prev Med. 1979 Jan;8(1):2-13. doi: 10.1016/0091-7435(79)90024-0. No abstract available. PMID 424377
- [Background] Borhani N: The Hypertension Detection and Follow-Up Program, in Onesti G and Klimt C (eds), Hypertension. Determinants, Complications, and Intervention, Grune & Stratton, New York, pp. 405-4l4, l979.
- [Background] Five-year findings of the hypertension detection and follow-up program. I. Reduction in mortality of persons with high blood pressure, including mild hypertension. Hypertension Detection and Follow-up Program Cooperative Group. JAMA. 1979 Dec 7;242(23):2562-71. PMID 490882
- [Background] Five-year findings of the hypertension detection and follow-up program. II. Mortality by race-sex and age. Hypertension Detection and Follow-up Program Cooperative Group. JAMA. 1979 Dec 7;242(23):2572-7. doi: 10.1001/jama.1979.03300230028022. PMID 490883
- [Background] Wassertheil-Smoller S, Apostolides A, Miller M, Oberman A, Thom T. Recent status of detection, treatment, and control of hypertension in the community. J Community Health. 1979 Winter;5(2):82-93. doi: 10.1007/BF01324010. PMID 262241
- [Background] Apostolides AY, Cutter G, Kraus JF, Oberman A, Blaszkowski T, Borhani NO, Entwisle G. Impact of hypertension information on high blood pressure control between 1973 and 1978. Hypertension. 1980 Sep-Oct;2(5):708-13. doi: 10.1161/01.hyp.2.5.708. PMID 7419272
- [Background] Cutter G, Heyden S, Kasteler J, Kraus JF, Lee ES, Shipley T, Stromer M. Mortality surveillance in collaborative trials. Am J Public Health. 1980 Apr;70(4):394-400. doi: 10.2105/ajph.70.4.394. PMID 7361958
- [Background] Cowan L, Detels R, Farber M, Lee ES, McCray G, O'Flynn S, Parnell MJ. Residential mobility and long-term treatment of hypertension. J Community Health. 1980 Spring;5(3):159-66. doi: 10.1007/BF01323988. PMID 7364958
- [Background] Stamler J, Borhani NO: Interview: HDFP Mortality and Morbidity. Hypertension Report, 1(l):l2-l4, l980.
- [Background] Stamler J: Clinical Ramifications of the Hypertension Detection and Follow-up Program: Benefits of Treatment Outweigh Risks. Symposia Reporter, 4(2):l2-l4, May l980.
- [Background] Langford HG: Clinical Ramifications of the Hypertension Detection and Follow-up Program: HDFP Methodology and Results: Overview. Symposia Reporter, 4(2):3-6, May l980.
- [Background] Borhani NO: Clinical Ramifications of the Hypertension Detection and Follow-up Program: SC Yields Lower Mortality and Morbidity. Symposia Reporter, 4(2):l6, May l980.
- [Background] Five-year findings of the hypertension detection and follow-up program. III. Reduction in stroke incidence among persons with high blood pressure. Hypertension Detection and Follow-up Program Cooperative Group. JAMA. 1982 Feb 5;247(5):633-8. PMID 7033578
- [Background] Apostolides AY, Cutter G, Daugherty SA, Detels R, Kraus J, Wassertheil-Smoller S, Ware J. Three-year incidence of hypertension in thirteen U.S. communities. On behalf of the Hypertension Detection and Follow-up Program cooperative group. Prev Med. 1982 Sep;11(5):487-99. doi: 10.1016/0091-7435(82)90063-9. No abstract available. PMID 7156059
- [Background] Kraus JF, Conley A, Hardy R, Sexton M, Sweezy Z. Relationship of demographic characteristics of interviewers to blood pressure measurements. J Community Health. 1982 Fall;8(1):3-12. doi: 10.1007/BF01324392. PMID 7186909
- [Background] Curb JD, Hardy RJ, Labarthe DR, Borhani NO, Taylor JO. Reserpine and breast cancer in the Hypertension Detection and Follow-Up Program. Hypertension. 1982 Mar-Apr;4(2):307-11. doi: 10.1161/01.hyp.4.2.307. PMID 7040229
- [Background] Shulman N, Cutter G, Daugherty R, Sexton M, Pauk G, Taylor MJ, Tyler M. Correlates of attendance and compliance in the hypertension detection and follow-up program. Control Clin Trials. 1982 Mar;3(1):13-27. doi: 10.1016/0197-2456(82)90016-2. PMID 7067470
- [Background] Smith EO, Curb JD, Hardy RJ, Hawkins CM, Tyroler HA. Clinic attendance in the hypertension detection and follow-up program. Hypertension. 1982 Sep-Oct;4(5):710-5. doi: 10.1161/01.hyp.4.5.710. No abstract available. PMID 7106938
- [Background] Curb JD, Ford C, Hawkins CM, Smith EO, Zimbaldi N, Carter B, Cooper C. A coordinating center in a clinical trial: the Hypertension Detection and Followup Program. Control Clin Trials. 1983 Sep;4(3):171-86. doi: 10.1016/0197-2456(83)90001-6. PMID 6641231
- [Background] Daugherty SA, Entwisle G, et al (Eds.): Hypertension Detection and Follow-Up Program: Baseline Characteristics of the Enumerated, Screened, and Hypertensive Participants. Hypertension (AHA Monograph No. 104), 1983.
- [Background] Hardy RJ, Hawkins CM. The impact of selected indices of antihypertensive treatment on all-cause mortality. Am J Epidemiol. 1983 May;117(5):566-74. doi: 10.1093/oxfordjournals.aje.a113579. PMID 6846314
- [Background] Morris DL, Borhani NO, Fitzsimons E, Hardy RJ, Hawkins CM, Kraus JF, Labarthe DR, Mastbaum L, Payne GH. Serum cholesterol and cancer in the Hypertension Detection and Follow-up Program. Cancer. 1983 Nov 1;52(9):1754-9. doi: 10.1002/1097-0142(19831101)52:93.0.co;2-j. PMID 6616425
- [Background] Willett WC, Polk BF, Morris JS, Stampfer MJ, Pressel S, Rosner B, Taylor JO, Schneider K, Hames CG. Prediagnostic serum selenium and risk of cancer. Lancet. 1983 Jul 16;2(8342):130-4. doi: 10.1016/s0140-6736(83)90116-2. PMID 6134981
- [Background] Tyroler HA: Race, Education and Five-Year Mortality In HDFP Stratum I Referred-care Males in Mild Hypertension: Recent Advances, Gross R and Strasser T (Eds). New York, Raven Press, 163- , 1983.
- [Background] Daugherty SA. Hypertension detection and follow-up program. Description of the enumerated and screened population. Hypertension. 1983 Nov-Dec;5(6 Pt 2):IV1-43. doi: 10.1161/01.hyp.5.6_pt_2.iv1. No abstract available. PMID 6360872
- [Background] Taylor JO, Borhani NO, Entwisle G, Farber M, Hawkins CM. Hypertension detection and follow-up program. Summary of the baseline characteristics of the hypertensive participants. Hypertension. 1983 Nov-Dec;5(6 Pt 2):IV44-50. doi: 10.1161/01.hyp.5.6_pt_2.iv44. No abstract available. PMID 6360875
- [Background] Kraus JF, Curb JD, Cutter G, Daugherty SA, Neill KC, Wassertheil-Smoller S. Hypertension detection and follow-up program. Baseline medical history characteristics of the hypertensive participants. Hypertension. 1983 Nov-Dec;5(6 Pt 2):IV51-91. doi: 10.1161/01.hyp.5.6_pt_2.iv51. No abstract available. PMID 6360876
- [Background] Polk BF, Cutter G, Daugherty RM, Gosch F, Heyden S, Shulman N, Tyroler HA. Hypertension detection and follow-up program. Baseline physical examination characteristics of the hypertensive participants. Hypertension. 1983 Nov-Dec;5(6 Pt 2):IV92-132. doi: 10.1161/01.hyp.5.6_pt_2.iv92. No abstract available. PMID 6360877
- [Background] Maxwell MH, Fitzsimmons E, Harrist R, Hotchkiss J, Langford HG, Payne GH, Schneider KA, Varaday P. Hypertension detection and follow-up program. Baseline laboratory examination characteristics of the hypertensive participants. Hypertension. 1983 Nov-Dec;5(6 Pt 2):IV133-59. doi: 10.1161/01.hyp.5.6_pt_2.iv133. No abstract available. PMID 6360873
- [Background] Prineas RJ, Castle CH, Curb JD, Harrist R, Lewin A, Stamler J. Hypertension detection and follow-up program. Baseline electrocardiographic characteristics of the hypertensive participants. Hypertension. 1983 Nov-Dec;5(6 Pt 2):IV160-89. doi: 10.1161/01.hyp.5.6_pt_2.iv160. No abstract available. PMID 6360874
- [Background] Oberman A, Blaufox MD, Entwisle G, Harrist R. Hypertension detection and follow-up program. Baseline chest radiographic characteristics of the hypertensive participants. Hypertension. 1983 Nov-Dec;5(6 Pt 2):IV190-200. doi: 10.1161/01.hyp.5.6_pt_2.iv190. No abstract available. PMID 6654456
- [Background] Polk BF, Harlan LC, Cooper SP, Stromer M, Ignatius J, Mull H, Blaszkowski TP. Disability days associated with detection and treatment in a hypertension control program. Am J Epidemiol. 1984 Jan;119(1):44-53. doi: 10.1093/oxfordjournals.aje.a113724. PMID 6691335
- [Background] Willett WC, Polk BF, Underwood BA, Stampfer MJ, Pressel S, Rosner B, Taylor JO, Schneider K, Hames CG. Relation of serum vitamins A and E and carotenoids to the risk of cancer. N Engl J Med. 1984 Feb 16;310(7):430-4. doi: 10.1056/NEJM198402163100705. PMID 6537988
- [Background] Langford HG, Oberman A, Borhani NO, Entwisle G, Tung B. Black-white comparison of indices of coronary heart disease and myocardial infarction in the stepped-care cohort of the Hypertension Detection and Follow-Up Program. Am Heart J. 1984 Sep;108(3 Pt 2):797-801. doi: 10.1016/0002-8703(84)90674-4. PMID 6475749
- [Background] The effect of antihypertensive drug treatment on mortality in the presence of resting electrocardiographic abnormalities at baseline: the HDFP experience. The Hypertension Detection and Follow-up Program Cooperative Research Group. Circulation. 1984 Dec;70(6):996-1003. doi: 10.1161/01.cir.70.6.996. PMID 6388901
- [Background] Five-year findings of the Hypertension Detection and Follow-up Program. Prevention and reversal of left ventricular hypertrophy with antihypertensive drug therapy. Hypertension Detection and Follow-up Program Cooperative Group. Hypertension. 1985 Jan-Feb;7(1):105-12. PMID 3156812
- [Background] Curb JD, Borhani NO, Blaszkowski TP, Zimbaldi N, Fotiu S, Williams W. Patient-perceived side effects to antihypertensive drugs. Am J Prev Med. 1985 Jan-Feb;1(1):36-40. PMID 3870892
- [Background] Curb JD, Borhani NO, Blaszkowski TP, Zimbaldi N, Fotiu S, Williams W. Long-term surveillance for adverse effects of antihypertensive drugs. JAMA. 1985 Jun 14;253(22):3263-8. PMID 3999311
- [Background] Effect of stepped care treatment on the incidence of myocardial infarction and angina pectoris. 5-Year findings of the hypertension detection and follow-up program. Hypertension. 1984 Mar-Apr;6(2 Pt 2):I198-206. doi: 10.1161/01.hyp.6.2_pt_2.i198. PMID 6724670
- [Background] Five-year findings of the Hypertension Detection and Follow-up Program: mortality by race-sex and blood pressure level. A further analysis. Hypertension Detection and Follow-up Program Cooperative Group. J Community Health. 1984 Summer;9(4):314-27. PMID 6480895
- [Background] Mortality findings for stepped-care and referred-care participants in the hypertension detection and follow-up program, stratified by other risk factors. The Hypertension Detection and Follow-up Program Cooperative Research Group. Prev Med. 1985 May;14(3):312-35. doi: 10.1016/0091-7435(85)90059-3. PMID 2865725
- [Background] Bell RL, Curb JD, Friedman LM, Payne GH. Termination of clinical trials: the beta-blocker heart attack trial and the hypertension detection and follow-up program experience. Control Clin Trials. 1985 Jun;6(2):102-11. doi: 10.1016/0197-2456(85)90115-1. PMID 4006483
- [Background] Lewin A, Blaufox MD, Castle H, Entwisle G, Langford H. Apparent prevalence of curable hypertension in the Hypertension Detection and Follow-up Program. Arch Intern Med. 1985 Mar;145(3):424-7. PMID 3872106
- [Background] Maxwell MH, Ford CE. Cardiovascular morbidity and mortality in HDFP patients 50-69 years old at entry. J Cardiovasc Pharmacol. 1985;7 Suppl 2:S5-9. doi: 10.1097/00005344-198507002-00002. PMID 2409370
- [Background] Heyden S, Borhani NO, Tyroler HA, Schneider KA, Langford HG, Hames CG, Hutchinson R, Oberman A. The relationship of weight change to changes in blood pressure, serum uric acid, cholesterol and glucose in the treatment of hypertension. J Chronic Dis. 1985;38(4):281-8. doi: 10.1016/0021-9681(85)90073-6. PMID 3889027
- [Background] Implications of the Hypertension Detection and Follow-up Program. The Hypertension Detection and Follow-up Program Cooperative Group. Prog Cardiovasc Dis. 1986 Nov-Dec;29(3 Suppl 1):3-10. doi: 10.1016/0033-0620(86)90031-9. No abstract available. PMID 3538179
- [Background] Davis BR, Ford CE, Remington RD, Stamler R, Hawkins CM. The Hypertension Detection and Follow-up Program design, methods, and baseline characteristics and blood pressure response of the study population. Prog Cardiovasc Dis. 1986 Nov-Dec;29(3 Suppl 1):11-28. doi: 10.1016/0033-0620(86)90032-0. No abstract available. PMID 3538177
- [Background] Langford HG, Stamler J, Wassertheil-Smoller S, Prineas RJ. All-cause mortality in the Hypertension Detection and Follow-up Program: findings for the whole cohort and for persons with less severe hypertension, with and without other traits related to risk of mortality. Prog Cardiovasc Dis. 1986 Nov-Dec;29(3 Suppl 1):29-54. doi: 10.1016/0033-0620(86)90033-2. No abstract available. PMID 3538178
- [Background] Borhani NO, Blaufox MD, Oberman A, Polk BF. Incidence of coronary heart disease and left ventricular hypertrophy in the Hypertension Detection and Follow-up Program. Prog Cardiovasc Dis. 1986 Nov-Dec;29(3 Suppl 1):55-62. doi: 10.1016/0033-0620(86)90034-4. No abstract available. PMID 2947267
- [Background] Daugherty SA, Berman R, Entwisle G, Haerer AF. Cerebrovascular events in the Hypertension Detection and Follow-up Program. Prog Cardiovasc Dis. 1986 Nov-Dec;29(3 Suppl 1):63-72. doi: 10.1016/0033-0620(86)90035-6. No abstract available. PMID 3538180
- [Background] Curb JD, Maxwell MH, Schneider KA, Taylor JO, Shulman NB. Adverse effects of antihypertensive medications in the Hypertension Detection and Follow-up Program. Prog Cardiovasc Dis. 1986 Nov-Dec;29(3 Suppl 1):73-88. doi: 10.1016/0033-0620(86)90036-8. No abstract available. PMID 3538181
- [Background] Cressman MD, Gifford RW Jr. Clinicians' interpretation of the results and implications of the Hypertension Detection and Follow-up Program. Prog Cardiovasc Dis. 1986 Nov-Dec;29(3 Suppl 1):89-97. doi: 10.1016/0033-0620(86)90037-x. No abstract available. PMID 3538182
- [Background] Abernethy J, Borhani NO, Hawkins CM, Crow R, Entwisle G, Jones JW, Maxwell MH, Langford H, Pressel S. Systolic blood pressure as an independent predictor of mortality in the Hypertension Detection and Follow-up Program. Am J Prev Med. 1986 May-Jun;2(3):123-32. PMID 3453169
- [Background] Harlan LC, Polk BF, Cooper S, Blaszkowski TP, Ignatius-Smith J, Stromer M, Mull H. Effects of labeling and treatment of hypertension on perceived health. Am J Prev Med. 1986 Sep-Oct;2(5):256-61. PMID 3453188
- [Background] Williams WR, Schneider KA, Borhani NO, Schnaper HW, Slotkoff LM, Ellefson RD. The relationship between diuretics and serum cholesterol in Hypertension Detection and Follow-up Program participants. Am J Prev Med. 1986 Sep-Oct;2(5):248-55. PMID 3453187
- [Background] Ford CE, Langford HG, Palmer MJ. Recruitment in the hypertension detection and follow-up program. Control Clin Trials. 1987 Dec;8(4 Suppl):54S-67S. doi: 10.1016/0197-2456(87)90007-9. PMID 3440390
- [Background] Davis BR, Langford HG, Blaufox MD, Curb JD, Polk BF, Shulman NB. The association of postural changes in systolic blood pressure and mortality in persons with hypertension: the Hypertension Detection and Follow-up Program experience. Circulation. 1987 Feb;75(2):340-6. doi: 10.1161/01.cir.75.2.340. PMID 3802437
- [Background] Educational level and 5-year all-cause mortality in the Hypertension Detection and Follow-up Program. Hypertension Detection and Follow-up Program Cooperative Group. Hypertension. 1987 Jun;9(6):641-6. PMID 3583404
- [Background] Curb JD, Schneider K, Taylor JO, Maxwell M, Shulman N. Antihypertensive drug side effects in the Hypertension Detection and Follow-up Program. Hypertension. 1988 Mar;11(3 Pt 2):II51-5. doi: 10.1161/01.hyp.11.3_pt_2.ii51. PMID 3350594
- [Background] Davis BR, Curb JD, Borhani NO, Prineas RJ, Molteni A. Coffee consumption and serum cholesterol in the hypertension detection and follow-up program. Am J Epidemiol. 1988 Jul;128(1):124-36. doi: 10.1093/oxfordjournals.aje.a114935. PMID 3381821
- [Background] Martin JB, Annegers JF, Curb JD, Heyden S, Howson C, Lee ES, Lee M. Mortality patterns among hypertensives by reported level of caffeine consumption. Prev Med. 1988 May;17(3):310-20. doi: 10.1016/0091-7435(88)90006-0. PMID 3043418
- [Background] Persistence of reduction in blood pressure and mortality of participants in the Hypertension Detection and Follow-up Program. Hypertension Detection and Follow-up Program Cooperative Group. JAMA. 1988 Apr 8;259(14):2113-22. PMID 3346988
- [Background] Cooper SP, Hardy RJ, Labarthe DR, Hawkins CM, Smith EO, Blaufox MD, Cooper CJ, Entwisle G, Maxwell MH. The relation between degree of blood pressure reduction and mortality among hypertensives in the Hypertension Detection and Follow-Up Program. Am J Epidemiol. 1988 Feb;127(2):387-403. doi: 10.1093/oxfordjournals.aje.a114812. PMID 3276167
- [Background] Daugherty SA. Mortality findings beyond five years in the hypertension detection and follow-up program (HDFP). J Hypertens Suppl. 1988 Dec;6(4):S597-601. doi: 10.1097/00004872-198812040-00187. PMID 3071594
- [Background] Shulman NB, Ford CE, Hall WD, Blaufox MD, Simon D, Langford HG, Schneider KA. Prognostic value of serum creatinine and effect of treatment of hypertension on renal function. Results from the hypertension detection and follow-up program. The Hypertension Detection and Follow-up Program Cooperative Group. Hypertension. 1989 May;13(5 Suppl):I80-93. doi: 10.1161/01.hyp.13.5_suppl.i80. PMID 2490833
- [Background] Stamler R, Ford CE, Stamler J. Why do lean hypertensives have higher mortality rates than other hypertensives? Findings of the Hypertension Detection and Follow-up Program. Hypertension. 1991 Apr;17(4):553-64. doi: 10.1161/01.hyp.17.4.553. PMID 2013482
- [Background] Finnerty FA Jr, Shaw LW, Himmelsbach CK. Hypertension in the inner city. II. Detection and follow-up. Circulation. 1973 Jan;47(1):76-8. doi: 10.1161/01.cir.47.1.76. No abstract available. PMID 4686606
- [Background] Hyden S, Tyroler HA, Hames CG, Bartel A, Thompson JW, Krishan I, Rosenthal T. Diet treatment of obese hypertensives. Clin Sci Mol Med Suppl. 1973 Aug;45 Suppl 1:209s-12. doi: 10.1042/cs045209s. No abstract available. PMID 4593567
- [Background] Labarthe DR, Hawkins CM, Remington RD. Evaluation of performance of selected devices for measuring blood pressure. Am J Cardiol. 1973 Sep 20;32(4):546-53. doi: 10.1016/s0002-9149(73)80046-3. No abstract available. PMID 4729723
- [Background] Apostolides A, Hebel JR, McDill MS, Henderson MM. High blood pressure: its care and consequences in urban centres. Int J Epidemiol. 1974 Jun;3(2):105-18. doi: 10.1093/ije/3.2.105. No abstract available. PMID 4277505
- [Background] Henderson M, Apostolides A, Entwisle G, Hebel R. A study of hypertension in a black urban community: preliminary epidemiologic findings. Prev Med. 1974 Sep;3(3):334-43. doi: 10.1016/0091-7435(74)90045-0. No abstract available. PMID 4411765
- [Background] Wassertheil-Smoller S, Bell B, Blaufox MD. Computer-aided management of hypertensive patients. Med Care. 1975 Dec;13(12):1044-54. doi: 10.1097/00005650-197512000-00006. PMID 1195905
- [Background] Wassertheil-Smoller S, Blaufox MD. Planning case-finding activities for a community hypertension-control program. Bull N Y Acad Med. 1976 Jul-Aug;52(6):648-56. No abstract available. PMID 1067879
- [Background] Langford HG, Watson RL, Thomas JG. Salt intake and the treatment of hypertension. Am Heart J. 1977 Apr;93(4):531-2. doi: 10.1016/s0002-8703(77)80418-3. No abstract available. PMID 842451
- [Background] Schlant RC, Felner JL, Heymsfield SB, Gilbert CA, Shulman NB, Tuttle EP, and Blumenstein BA: Echocardiography and Essential Hypertension. Cardiovascular Medicine, 2:477-490, l977.
- [Background] Entwisle G, Apostolides AY, Hebel JR, Henderson MM. Target organ damage in black hypertensives. Circulation. 1977 May;55(5):792-6. doi: 10.1161/01.cir.55.5.792. PMID 139214
- [Background] Apostolides AY, Entwisle G, Ouellet R, Hebel JR. Improving trend in hypertension control in a black inner city community. Am J Epidemiol. 1978 Feb;107(2):113-9. doi: 10.1093/oxfordjournals.aje.a112513. PMID 623094
- [Background] Stamler R, Gosch FC, Stamler J, Lindberg HA, Hilker RR. A hypertension control program based on the workplace. Report on the Chicago Center. J Occup Med. 1978 Sep;20(9):618-25. doi: 10.1097/00043764-197809000-00010. PMID 702219
- [Background] Blaufox MD, Wassertheil-Smoller S. Improving blood pressure normalization. Follow-up of hypertension screening and methodologies. N Y State J Med. 1979 Feb;79(2):231-5. No abstract available. PMID 285353
- [Background] Ouellet RP, Apostolides AY, Entwisle G, Hebel JR. Estimated community impact of hypertension control in a high risk population. Am J Epidemiol. 1979 May;109(5):531-8. doi: 10.1093/oxfordjournals.aje.a112711. No abstract available. PMID 453176
- [Background] Smith EO, Hardy RJ, Cutter GR, Curb JD, and Hawkins CM: Application of Survival Analysis Techniques to Evaluation of Factors Affecting Compliance in a Clinical Trial of Hypertension Control. Controlled Clin Trials, l:59-69, l980.
- [Background] Smith EO, Hardy RJ, Cutter GR. A two-compartment regression model applied to compliance in a hypertension treatment program. J Chronic Dis. 1980;33(10):645-51. doi: 10.1016/0021-9681(80)90007-7. No abstract available. PMID 7410524
- [Background] Smith EO, Hardy RJ, Cooper CJ, Hawkins CM. Two-compartment Markov regression analysis. Comput Programs Biomed. 1980 Dec;12(2-3):129-40. doi: 10.1016/0010-468x(80)90059-8. PMID 7249589
- [Background] The hypertension detection and follow-up program: Hypertension detection and follow-up program cooperative group. Prev Med. 1976 Jun;5(2):207-15. doi: 10.1016/0091-7435(76)90039-6. No abstract available. PMID 935073
- [Background] Blood pressure studies in 14 communities. A two-stage screen for hypertension. JAMA. 1977 May 30;237(22):2385-91. doi: 10.1001/jama.1977.03270490025018. PMID 576938
- [Background] Taylor J. The hypertension detection and follow-up program: a progress report. Circ Res. 1977 May;40(5 Suppl 1):I106-9. PMID 576851
- [Background] Langford HG. Further analyses of the hypertension detection and follow-up program. Drugs. 1986;31 Suppl 1:23-8. doi: 10.2165/00003495-198600311-00006. PMID 2941267
- [Background] Race, education and prevalence of hypertension. Am J Epidemiol. 1977 Nov;106(5):351-61. PMID 920724
- Available data/document: Individual Participant Data Set: HDFP — http://biolincc.nhlbi.nih.gov/studies/hdfp/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/hdfp/